CLINICAL TRIAL: NCT05659147
Title: Imaging Biomarkers of Pancreatic Function and Disease
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-0779; R01DK132346 (NIH)
Record Dates: First submitted 2022-11-22; First posted 2022-12-21 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Pancreatitis; Diabetes Mellitus
Keywords: MRI
MeSH Terms: conditions — Pancreatitis; Diabetes Mellitus | interventions — Hematologic Tests; Occult Blood; Secretin

STUDY DESIGN:
Intervention Model Description: Participants will be prospectively recruited to one or more of four prospective imaging aims (Aims 1-4). All participants who enroll in any imaging Aim will have their images used for Aim 5 (image analysis aim) which will also include a retrospective component.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (5):
- Imaging markers of exocrine and endocrine insufficiency (Experimental): We will prospectively enroll 85 participants; 40 with known or suspected EPI and 45 controls (no known organic gastrointestinal pathology and no history of pancreatic disease) in this aim.
  Participants will be undergoing clinically-indicated endoscopy and will have endoscopic pancreatic function tests (ePFTs) collected for research during the clinically-indicated endoscopy examination. A research blood draw and a research stool collection will also be collected from all participants. Participants will undergo a research MRI examination with administration of intravenous secretin within 2 weeks of their clinical endoscopy but no sooner than 2 hours before or after endoscopy.
  Interventions: Diagnostic Test: Research MRI with administration of intravenous secretin; Diagnostic Test: Blood Tests; Diagnostic Test: Stool Tests; Other: Survey Completion; Diagnostic Test: Endoscopic pancreatic function tests (ePFTs); Drug: Secretin
- Imaging markers of diabetes and prediction of progression to diabetes (Experimental): We will prospectively enroll 30 participants; 10 with a single episode of acute pancreatitis, 10 with acute recurrent pancreatitis, and 10 with pancreatitis-related diabetes in this aim.
  Participants will undergo a research MRI examination. Participants will also undergo a research blood draw for laboratory analysis and to enable gene sequencing for gene mutations associated with heritable pancreatitis. We will assess the association between identified gene variants and the presence of diabetes and will construct models based on identified variants to predict progression to diabetes.
  Interventions: Diagnostic Test: Research MRI without administration of intravenous secretin; Genetic: Genetic Sequencing; Diagnostic Test: Blood Tests; Other: Survey Completion
- Imaging stratification of stages of pancreatitis (Experimental): We will prospectively enroll 60 participants; 15 healthy controls, 15 participants with a single episode of acute pancreatitis, 15 participants with acute recurrent pancreatitis, and 15 participants with chronic pancreatitis.
  A research blood draw and a research stool collection will be collected from all participants. Participants will undergo a research MRI examination with administration of intravenous secretin.
  Interventions: Diagnostic Test: Research MRI with administration of intravenous secretin; Diagnostic Test: Blood Tests; Diagnostic Test: Stool Tests; Other: Survey Completion; Drug: Secretin
- Imaging reproducibility (Experimental): We will prospectively enroll up to 20 participants enrolled in Aims 1 or 3 (up to 5 controls and 15 patients with pancreatic disease) to undergo repeat research MRI imaging between 24 hours and 14 days after their first research MRI.
  Participants will undergo a research MRI examination with administration of intravenous secretin, identical to the research MRI performed under Aims 1 or 3. MRI images will be quantitatively analyzed and agreement between the two MRI examinations (1st and repeat MRI) will be assessed.
  Interventions: Diagnostic Test: Research MRI with administration of intravenous secretin; Drug: Secretin
- Automated or semi-automated image analysis (No Intervention): We will use images prospectively collected under Aims 1-3, as well as existing images that had been obtained for clinical care of children with pancreatitis at CCHMC to develop and optimize image processing pipelines for MRI images. Performance of these pipelines will be benchmarked against manual segmentation performed by multiple observers.

INTERVENTIONS:
Diagnostic Test: Research MRI without administration of intravenous secretin — Participants will undergo a research MRI examination. MRI images will be quantitatively analyzed and will be compared to / used to predict diabetes.
  Arms: Imaging markers of diabetes and prediction of progression to diabetes
Diagnostic Test: Research MRI with administration of intravenous secretin — Participants will undergo a research MRI examination with intravenous administration of secretin. MRI images will be quantitatively analyzed and will be compared to / used to predict exocrine and endocrine pancreatic insufficiency based on the reference standards of ePFTs or fecal elastase and blood hemoglobin A1c (HbA1c) and fasting glucose, respectively.
  Arms: Imaging markers of exocrine and endocrine insufficiency; Imaging reproducibility; Imaging stratification of stages of pancreatitis
Genetic: Genetic Sequencing — Blood will be drawn to enable gene sequencing for gene mutations associated with heritable pancreatitis. We will assess the association between identified gene variants and the presence of diabetes and will construct models based on identified variants to predict progression to diabetes.
  Arms: Imaging markers of diabetes and prediction of progression to diabetes
Diagnostic Test: Blood Tests — Research blood draw (for markers of pancreatic endocrine insufficiency)
  Arms: Imaging markers of diabetes and prediction of progression to diabetes; Imaging markers of exocrine and endocrine insufficiency; Imaging stratification of stages of pancreatitis
Diagnostic Test: Stool Tests — Research stool collection (for fecal elastase as a marker of exocrine insufficiency)
  Arms: Imaging markers of exocrine and endocrine insufficiency; Imaging stratification of stages of pancreatitis
Other: Survey Completion — Participants will be contacted to complete a survey and their charts will be reviewed annually after research MRI to identify any evidence of subsequent development of pancreatic endocrine insufficiency or progression of pancreatitis. Survey and chart review will occur within +/- 14 days of the anniversary date.
  Arms: Imaging markers of diabetes and prediction of progression to diabetes; Imaging markers of exocrine and endocrine insufficiency; Imaging stratification of stages of pancreatitis
Diagnostic Test: Endoscopic pancreatic function tests (ePFTs) — At least two duodenal fluid aspirates will be collected over 15 minutes following secretin administration. Aspirates will be immediately pH tested and will be submitted for analysis of bicarbonate, enzyme (trypsin, amylase, lipase, chymotrypsin) activity, and total protein.
  Arms: Imaging markers of exocrine and endocrine insufficiency
Drug: Secretin — Participants enrolled in Aim 1, Aim 3, and Aim 4 will receive intravenous secretin at a dose of 0.2 mcg/kg (maximum 16 mcg).
  Participants in Aim 1 will receive two doses (1 during endoscopy and 1 during MRI). Participants in Aim 3 will receive one dose during MRI.
  Participants in Aim 4 will receive two doses (1 during each MRI).
  Secretin for intravenous use is FDA-approved for stimulation of pancreatic secretions, including bicarbonate, to aid in the diagnosis of exocrine pancreas dysfunction. Safety and effectiveness of secretin in pediatrics have not been established. However, secretin is routinely used in children at CCHMC at the same dose at which it will be administered for this study.
  Arms: Imaging markers of exocrine and endocrine insufficiency; Imaging reproducibility; Imaging stratification of stages of pancreatitis

SUMMARY:
This study seeks to understand the performance of MRI to characterize pancreatitis and predict chronic complications (endocrine and exocrine) of pancreatitis. Through multiple aims, the investigators will benchmark MRI against relevant reference standards (e.g. endoscopic pancreatic function tests, laboratory data). The investigators will also characterize repeatability of the imaging findings and will work to develop methods to simplify and automate analysis of the MRI images.

Research interventions depend on the Aim(s) participants enroll in but include: endoscopic pancreatic function testing (added on to clinically indicated upper GI endoscopy), blood tests, stool tests, gene sequencing, and survey completion. All participants will undergo research MRI examinations, a subset of which will include administration of intravenous secretin.

DETAILED DESCRIPTION:
Pancreatitis can be acute [AP], acute recurrent [ARP] (defined as two discrete attacks with interval resolution), or chronic [CP]. Adult studies show that up to 40% of patients develop abnormal glucose metabolism after a single attack of AP, with a 2.5x increased risk of diabetes. CP is defined, in part, by the presence of established endocrine (diabetes) or exocrine pancreatic insufficiency [EPI]. Currently, it is not possible to non-invasively diagnose or predict development of pancreatitis-related endocrine or exocrine insufficiency.

The investigator's data has shown that CFTR gene variants play a significant role in progression to diabetes post first attack AP. Existing literature suggests that imaging findings such as decreased pancreas volume are associated with diabetes, but this has not been systematically studied in children.

EPI, defined as insufficient secretion of digestive enzymes and fluid by the pancreas, can have significant effects in childhood including malnutrition, osteoporosis, and growth failure. If diagnosed early, EPI can be treated with pancreatic enzyme replacement, improving nutrition and stabilizing growth. Unfortunately, diagnosing EPI early and accurately is a challenge in children and it is currently not possible to predict progression to CP or development of EPI.

Magnetic resonance imaging (MRI) is a powerful, non-invasive technique, capable of characterizing pancreatic disease. Quantitative non-contrast MRI techniques are attractive as potential markers of pancreatic disease but they have not been validated for diagnosis or prediction of diabetes or EPI in children and they have not been explored for staging of pediatric pancreatitis.

The overall goals of this study are to:

1. Define associations between non-invasive, quantitative MRI measures and established measures of pancreas health and function including diabetes and EPI in children
2. Identify clinical, genetic and imaging-related factors that predict progression to diabetes in children with pancreatitis.

ELIGIBILITY:
Aim 1-

Patient Group:

Inclusion Criteria:

* Age 5 to <21 years
* Scheduled for clinically-indicated gastrointestinal endoscopy
* Clinical diagnosis or suspicion of exocrine pancreatic insufficiency

Exclusion Criteria:

* Complete fatty replacement of pancreas on prior imaging
* Current acute pancreatitis or acute pancreatitis less than 30 days prior to research MRI
* Need for sedation for MRI
* Contraindication to MRI (implanted metal hardware)
* Allergy to secretin
* Pregnancy

Control Group:

Inclusion Criteria:

* Age 5 to <21 years
* Scheduled for clinically-indicated gastrointestinal endoscopy

Exclusion Criteria:

* Sweat chloride >60 mmol/L
* Clinical diagnosis of gastrointestinal pathology
* Clinical diagnosis or history of pancreatic disease
* Complete fatty replacement of pancreas on prior imaging
* Current acute pancreatitis or acute pancreatitis less than 30 days prior to research MRI
* Need for sedation for MRI
* Contraindication to MRI (implanted metal hardware)
* Allergy to secretin
* Pregnancy

Aim 2-

Acute Pancreatitis Group:

Inclusion Criteria:

* Age 5 to <21 years
* Clinically documented episode of acute pancreatitis

Exclusion Criteria:

* More than one episode of acute pancreatitis
* Current acute pancreatitis or acute pancreatitis less than 30 days prior to research MRI
* Need for sedation for MRI
* Contraindication to MRI (implanted metal hardware)
* Pregnancy

Acute Recurrent Pancreatitis Group:

Inclusion Criteria:

* Age 5 to <21 years
* Clinical diagnosis of acute recurrent pancreatitis

Exclusion Criteria:

* Current acute pancreatitis or acute pancreatitis less than 30 days prior to research MRI
* Need for sedation for MRI
* Contraindication to MRI (implanted metal hardware)
* Pregnancy

Pancreatitis-Related Diabetes Group:

Inclusion Criteria:

* Age 5 to <21 years
* Clinical diagnosis of pancreatitis-related diabetes

Exclusion Criteria:

* Current acute pancreatitis or acute pancreatitis less than 30 days prior to research MRI
* Need for sedation for MRI
* Contraindication to MRI (implanted metal hardware)
* Pregnancy

Aim 3-

Control Group:

Inclusion Criteria:

• Age 5 to <21 years

Exclusion Criteria:

* Sweat chloride >60 mmol/L
* Clinical diagnosis of gastrointestinal pathology
* Clinical diagnosis or history of pancreatic disease, including acute pancreatitis
* Need for sedation for MRI
* Contraindication to MRI (implanted metal hardware)
* Allergy to secretin
* Pregnancy

Acute Pancreatitis Group:

Inclusion Criteria:

* Age 5 to <21 years
* Clinically documented episode of acute pancreatitis

Exclusion Criteria:

* More than one episode of acute pancreatitis
* Current acute pancreatitis or acute pancreatitis less than 30 days prior to research MRI
* Need for sedation for MRI
* Contraindication to MRI (implanted metal hardware)
* Allergy to secretin
* Pregnancy

Acute Recurrent Pancreatitis Group:

Inclusion Criteria:

* Age 5 to <21 years
* Clinical diagnosis of acute recurrent pancreatitis with no evidence of CP or EPI

Exclusion Criteria:

* Current acute pancreatitis or acute pancreatitis less than 30 days prior to research MRI
* Need for sedation for MRI
* Contraindication to MRI (implanted metal hardware)
* Allergy to secretin
* Pregnancy

Chronic Pancreatitis Group:

Inclusion Criteria:

* Age 5 to <21 years
* Clinical diagnosis of chronic pancreatitis

Exclusion Criteria:

* Current acute pancreatitis or acute pancreatitis less than 30 days prior to research MRI
* Need for sedation for MRI
* Contraindication to MRI (implanted metal hardware)
* Allergy to secretin
* Pregnancy

Aim 4-

Inclusion Criteria:

* Age 5 to <21 years
* Completed research MRI under Aims 1 or 3 of this study

Exclusion Criteria:

* Failed/unable to complete first research MRI under Aims 1 or 3
* Episode of acute pancreatitis since first research MRI
* Current acute pancreatitis
* Any gastrointestinal surgery or pancreas intervention (e.g. ERCP) since first research MRI
* Need for sedation for MRI
* Contraindication to MRI (implanted metal hardware)
* Allergy to secretin
* Pregnancy

Aim 5-

Inclusion Criteria:

• MRI performed at CCHMC

Exclusion Criteria:

* Severe image artifact compromising image quality (judgement of study team)
* Age >21 years

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 195 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Pancreas volume as a predictor of pancreas health and function (including endocrine and exocrine pancreatic insufficiency). | 5 years
  2 x 2 table analyses of pancreas volume (categorized as normal vs. abnormal) vs. exocrine function (categorized as normal vs. abnormal)
Pancreas volume as a predictor of pancreas health and function (including endocrine and exocrine pancreatic insufficiency). | 5 years
  2 x 2 table analyses of pancreas volume (categorized as normal vs. abnormal) vs. endocrine function (categorized as normal vs. abnormal)
Pancreas T1 signal as a predictor of pancreas health and function (including endocrine and exocrine pancreatic insufficiency). | 5 years
  2 x 2 table analyses of pancreas T1 signal (categorized as normal vs. abnormal) vs. exocrine function (categorized as normal vs. abnormal)
Pancreas T1 signal as a predictor of pancreas health and function (including endocrine and exocrine pancreatic insufficiency). | 5 years
  2 x 2 table analyses of pancreas T1 signal intensity (categorized as normal vs. abnormal) vs. endocrine function (categorized as normal vs. abnormal)
Pancreas secreted fluid volume as a predictor of pancreas health and function (including endocrine and exocrine pancreatic insufficiency). | 5 years
  2 x 2 table analyses of pancreas secreted fluid volume (categorized as normal vs. abnormal) vs. exocrine function (categorized as normal vs. abnormal)
Pancreas secreted fluid volume as a predictor of pancreas health and function (including endocrine and exocrine pancreatic insufficiency). | 5 years
  2 x 2 table analyses of pancreas secreted fluid volume (categorized as normal vs. abnormal) vs. endocrine function (categorized as normal vs. abnormal)
Frequency of genetic mutations in patients progressing to diabetes vs. those not | 5 years
  Frequency of genetic mutations in each study group will be compared using 2x2 tables to identify mutations associated with development of diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Trout, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-12-02): https://cdn.clinicaltrials.gov/large-docs/47/NCT05659147/ICF_000.pdf